CLINICAL TRIAL: NCT05448924
Title: Isolated Growth Hormone Deficiency and Amennorrhea: Case Report
Brief Title: Isolated Growth Hormone Deficiency and Amennorrhea
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: OBGY-202206.04
Record Dates: First submitted 2022-06-26; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Growth Hormone Deficiency
Keywords: ISOLATED GROWTH HORMONE DEFICIENCY; AMENORRHEA
MeSH Terms: conditions — Dwarfism, Pituitary; Amenorrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hormone panel tests — Patient was subjected to a battery of hormone tests, including FSH, LH, estrogen, progesterone and growth hormone

SUMMARY:
This is a case report of a 14-year old female with no menstruation history.

DETAILED DESCRIPTION:
This is a case report of a 14-year-old with a chief complaint of inability to menstruate. Lab tests were done.

ELIGIBILITY:
Inclusion Criteria:

* A single female participant with amenorrhea

Exclusion Criteria:

* The study only included the above subject

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This 14-year old female came to the gynaecology clinic with a chief complaint of amenorrhea
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Growth hormone levels | 1 month after testing
  Growth hormone levels assessed by hormone panel

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Universitas Padjadjaran, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous patient data may be shared with reasonable written request to the authors

REFERENCES:
- [Background] Crottaz B, Uske A, Reymond MJ, Rey F, Temler E, Germond M, Gomez F. Normogonadotropic primary amenorrhea in a growth hormone-deficient woman with ectopic posterior pituitary: gonadotropin pulsatility and follicle-stimulating hormone bioactivity. J Endocrinol Invest. 1996 Jan;19(1):48-53. doi: 10.1007/BF03347858. PMID 8851692